CLINICAL TRIAL: NCT02231658
Title: Effects of Victoza® (Liraglutide) Versus Lyxumia® (Lixisenatide) on Gastroesophageal Reflux, Gastric Emptying and Gastric Acid Secretion
Brief Title: Effects of Victoza® Versus Lyxumia® on Gastroesophageal Reflux, Gastric Emptying and Gastric Acid Secretion
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Too challenging to recruit appropriate participants at an acceptable speed.
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GI-Motil
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide; lixisenatide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental): The highest injected once daily dose will be 1.8 mg s.c. for liraglutide.
  Interventions: Drug: Liraglutide
- Lixisenatide (Experimental): The highest injected once daily dose will be 20µg s.c. for lixisenatide.
  Interventions: Drug: Lixisenatide

INTERVENTIONS:
Drug: Liraglutide
  Arms: Liraglutide
Drug: Lixisenatide
  Arms: Lixisenatide

SUMMARY:
The present study will compare lixisenatide and liraglutide in a population of subjects with T2DM not optimally controlled on OADs and / or insulin, which is the target population for these medications.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male or female aged 18-65 years (both inclusive)
* T2DM diagnosis

Exclusion Criteria:

* Contraindications (including known or suspected hypersensitivity) to GLP-1 mimetics
* Use of GLP-1 mimetics or DPP-IV inhibitors
* Clinically relevant dysglycaemia as indicated by HbA1C ≥ 10%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline (week -1) in the number of reflux episodes | 24 hours after 10 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline (week -1) in the time of pH < 4.0 in the lower third of the oesophagus | After 10 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Juris Meier, MD, Principal Investigator — St. Josef Hospital Bochum
Locations (2):
- Germany (2):
  - St. Josef-Hospital, Universitätsklinik, Bochum
  - Profil Institut für Stoffwechselforschung GmbH, Neuss

REFERENCES:
- [Derived] Quast DR, Schenker N, Menge BA, Nauck MA, Kapitza C, Meier JJ. Effects of Lixisenatide Versus Liraglutide (Short- and Long-Acting GLP-1 Receptor Agonists) on Esophageal and Gastric Function in Patients With Type 2 Diabetes. Diabetes Care. 2020 Sep;43(9):2137-2145. doi: 10.2337/dc20-0720. Epub 2020 Jul 9. PMID 32647054